CLINICAL TRIAL: NCT00780598
Title: The OPAL Study: A Phase II Study to Evaluate the Efficacy, Safety and Tolerability of Tosedostat (CHR-2797) in Elderly Subjects With Treatment Refractory or Relapsed Acute Myeloid Leukemia
Brief Title: Safety and Anti-Disease Activity of Oral Tosedostat (CHR-2797) in Elderly Subjects With Refractory or Relapsed AML
Acronym: OPAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chroma Therapeutics (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHR-2797-038
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-03

CONDITIONS: Acute Myeloid Leukemia; AML
Keywords: Acute Myeloid Leukemia; AML; Cancer; Hematological malignancies; Elderly; Refractory; Relapsed; Blood disorder
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms; Hematologic Neoplasms; Recurrence; Hematologic Diseases | interventions — tosedostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tosedostat (Experimental): oral, once daily administration of tosedostat to evaluate its efficacy, safety and tolerability
  Interventions: Drug: Tosedostat

INTERVENTIONS:
Drug: Tosedostat — In Part A, approximately 70 subjects will be randomized to one of 2 dose regimens of tosedostat which will be administered orally, once daily. The dose regimens of tosedostat will be:
  * 120 mg for 6 months once daily, OR
  * 240 mg (induction dose) once daily for 2 months, followed by 120 mg(maintenance dose) for 4 months
  In Part B a further 130 subjects will receive the dose regimen of tosedostat identified in Part A as being appropriate, based on the interim analysis during Part A.
  Other Names: - CHR-2797; - Aminopeptidase inhibitor

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of tosedostat in elderly patients suffering from refractory or relapsed AML.

DETAILED DESCRIPTION:
There is an urgent need for novel compounds and treatment strategies for elderly patients with AML, particularly those with refractory or relapsed disease for whom there are few effective treatment options. Treatment options for elderly patients are further limited by co-morbidity and tolerability constraints.

Tosedostat is a new aminopeptidase inhibitor, which in preclinical experiments has shown potent activity in both in vitro and in vivo cancer models as a single agent. In early clinical studies particularly good results have been observed in refractory and relapsed AML in older patients and these observations form the basis for the current study.

This multi-center, open label phase II study will enrol approximately 70 subjects in Part A and 130 subjects in Part B.

ELIGIBILITY:
INCLUSION:

1. Signed, informed consent prior to any study specific procedure
2. Subjects with a confirmed diagnosis of AML according to WHO classification (excluding APL) who have had either a first CR lasting less than 12 months, or have not had a first CR and who will receive their first salvage therapy in this study [6]. For the purposes of this study, the following considerations apply:

   1. Subjects should have received only 1 induction course, but this may have consisted of more than one cycle of treatment, with different agents or doses in each cycle
   2. Induction courses should normally have consisted of agents and doses considered as standard of care for induction at the investigational site concerned
   3. Subjects may have received consolidation for any number of cycles. Consolidation will be considered as any regimens given while the subject was in remission
   4. Subjects who received hematopoietic stem cell transplant in first remission are eligible provided there has been no chemotherapy or other targeted therapies to treat a relapse, and there is no evidence of Graft Versus Host Disease (GVHD). Donor leukocyte infusion is allowed provided there is no evidence of hematologic relapse as defined by the International Working Group (IWG) [12]
3. Subject's peripheral blast count does not exceed 30,000/microlitre before randomization into the study. Hydroxyurea treatment or leukapheresis may be used prior to or during the screening period to achieve this - see Section 6.7.2.
4. Subject's life expectancy at randomization is judged to be at least 3 months
5. Subjects should have recovered from the adverse effects of prior therapies to grade ≤1 (according to CTCAE v3) (excluding alopecia and any adverse effects that are expected to be chronic and stable)
6. Subjects must have had a bone marrow aspiration performed within 28 days prior to randomization showing the subject has at least 5% blasts and is therefore neither in CR nor CRp. This may be done at the Screening Visit if appropriate and feasible
7. Subjects must have adequate hepatic and renal function including the following:

   1. Total bilirubin ≤ 1.5 x upper limit of normal (in the absence of Gilbert's syndrome)
   2. AST and ALT ≤ 2.5 x upper limit of normal
   3. Serum creatinine ≤ 1.5 x upper limit of normal
8. Age ≥ 60 years
9. Performance status ≤ 2 (ECOG scale)
10. Screening left ventricular ejection fraction (LVEF) ≥ 50%
11. Subject is able to comply with all study procedures during the study including all visits and tests
12. Male subjects with female partners of reproductive potential must use acceptable contraceptive methods for the duration of time on study and continue to do so for a further 3 months after the end of tosedostat treatment

Exclusion:

1. Subjects who have received prior therapy for first relapse or refractory disease (a second induction cycle within a single induction regimen is allowed as defined above in Inclusion criterion 2)
2. Anti-cancer therapy including chemotherapy, radiotherapy, endocrine therapy, immunotherapy or use of any other investigational agents within 2 weeks prior to randomization (with the exception of hydroxyurea which can be used in certain circumstances. Section 6.7.2)
3. Subjects with APL (FAB type M3) or CML in blast crisis
4. Any prior or co-existing medical condition that in the Investigator's judgment will substantially increase the risk associated with the subject's participation in the study
5. Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary study procedures
6. Significant* cardiovascular disease defined as:

   1. Congestive heart failure NYHA class 4
   2. Unstable angina pectoris
   3. History of myocardial infarction within 6 months prior to study entry
   4. Presence of clinically significant valvular heart disease
   5. Uncontrolled or clinically significant ventricular arrhythmia
   6. Presence of clinically significant conduction defect on screening ECG
   7. Uncontrolled hypertension (i.e., systolic BP >160mmHg, diastolic >90 mmHg in repeated measurements) despite adequate therapy
   8. Clinically significant atrial fibrillation *Grade 3/4 in the CTCAE v3 grading would generally be considered clinically significant, although this remains a judgment for the Investigator to make.
7. Gastrointestinal disorders that may interfere with absorption of drug
8. Active serious infection or sepsis at randomization
9. Clinically significant interstitial lung disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to evaluate the efficacy of tosedostat in elderly subjects with treatment refractory or relapsed AML by measuring CR and CRp. | Months 1, 2, 3 & 6

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of tosedostat in elderly subjects with treatment refractory or relapsed AML | Screening, Days 1, 2, 8, 15, 29, monthly thereafter + unschedulded visits when deemed necessary
To evaluate the efficacy of tosedostat in elderly subjects with treatment refractory or relapsed AML, as determined by measures other than CR and CRp for the type and duration of response | Months 1, 2, 3 & 6

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center; Karen Yee, MD, Principal Investigator — Princess Margaret Hospital, Canada; Eric Feldman, MD, Principal Investigator — Weill Cornell Medical College - New York Presbyterian Hospital; David Rizzieri, MD, Principal Investigator — Duke University; Joseph Jurcic, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Richard Larson, MD, Principal Investigator — University of Chicago; Hanna J Khoury, MD, Principal Investigator — Emory University Clinic; Harry Erba, MD, Principal Investigator — University of Michigan; Samir Parekh, MD, Principal Investigator — Montefiore Medical Center; Aarthi Shenoy, MD, Principal Investigator — Medstar Health Research Institute; Anjali Advani, MD, Principal Investigator — Taussig Cancer Institute; Shambavi Richard, MD, Principal Investigator — Stony Brook University Medical Center; Steven Allen, MD, Principal Investigator — Monter Cancer Center; Ehab Attalah, MD, Principal Investigator — Froedtert Hospital; John Storring, MD, Principal Investigator — Royal Victoria Hospital, Belfast; Gerrit J Ossenkoppele, MD, Principal Investigator — VUMC; Pieter Sonneveld, MD, Principal Investigator — Erasmus Medical Center; Gary Schiller, MD, Principal Investigator — UCLA Division of Hematology/oncology, Los Angeles; Peter Westervelt, MD, Principal Investigator — Washington University School of Medicine; Julio Hajdenberg, MD, Principal Investigator — MD Anderson Cancer centre, Orlando, FL; Stuart Goldberg, MD, Principal Investigator — John Theurer Cancer Center, Hackensack NJ
Locations (21):
- United States (17):
  - UCLA School of Medicine, Los Angeles, California
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - M.D. Anderson Cancer Center Orlando, Orlando, Florida
  - Emory University Clinic, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Michigan Health System, Ann Arbor, Michigan
  - Washington University, Oncology/Bone Marrow Transplant, St Louis, Missouri
  - John Theurer Cancer Center, Hackensack University Medical Center,, Hackensack, New Jersey
  - Monter Cancer Center, Lake Success, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College - New York Presbyterian Hospital, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center Weiler Division, The Bronx, New York
  - Duke Univeristy Medical Center, Durham, North Carolina
  - Taussig Cancer Institute, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Froedtert Hospital, Milwaukee, Wisconsin
- Canada (2):
  - Princess Margaret Hopsital, Toronto, Ontario
  - Royal Victoria Hospital, Montreal, Quebec
- Netherlands (2):
  - VUMC, Amsterdam
  - Erasmus MC, Rotterdam

REFERENCES:
- [Background] Krige D, Needham LA, Bawden LJ, Flores N, Farmer H, Miles LE, Stone E, Callaghan J, Chandler S, Clark VL, Kirwin-Jones P, Legris V, Owen J, Patel T, Wood S, Box G, Laber D, Odedra R, Wright A, Wood LM, Eccles SA, Bone EA, Ayscough A, Drummond AH. CHR-2797: an antiproliferative aminopeptidase inhibitor that leads to amino acid deprivation in human leukemic cells. Cancer Res. 2008 Aug 15;68(16):6669-79. doi: 10.1158/0008-5472.CAN-07-6627. PMID 18701491
- [Background] Estey E, Kornblau S, Pierce S, Kantarjian H, Beran M, Keating M. A stratification system for evaluating and selecting therapies in patients with relapsed or primary refractory acute myelogenous leukemia. Blood. 1996 Jul 15;88(2):756. No abstract available. PMID 8695828
- [Derived] Cortes J, Feldman E, Yee K, Rizzieri D, Advani AS, Charman A, Spruyt R, Toal M, Kantarjian H. Two dosing regimens of tosedostat in elderly patients with relapsed or refractory acute myeloid leukaemia (OPAL): a randomised open-label phase 2 study. Lancet Oncol. 2013 Apr;14(4):354-62. doi: 10.1016/S1470-2045(13)70037-8. Epub 2013 Feb 28. PMID 23453583